CLINICAL TRIAL: NCT01229644
Title: A Phase II Study of Crenolanib (CP-868,596), a Selective and Potent Inhibitor of PDGFR, for the Treatment of Adult Gliomas
Brief Title: Study of Crenolanib, a Selective and Potent Inhibitor of PDGFR, for the Treatment of Adult Gliomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-BRE-001
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Glioma
Keywords: Glioma; Brain Cancer; Recurrent glioma; Low grade glioma; PDGFR Inhibitor; Crenolanib (CP-868,596); Neo-adjuvant Therapy
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — crenolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): Adult newly diagnosed glioma (both low and high grade) patients, who are able to to take Crenolanib (CP-868,596) for at least 3 days prior to surgical resection.
  Interventions: Drug: Crenolanib (CP-868,596)
- Cohort B (Experimental): Adult patients with recurrent high grade glioma, including patients treated with bevacizumab. Patients are treated with Crenolanib (CP-868,596) continuously until they fulfill one of the criteria for study discontinuation.
  Interventions: Drug: Crenolanib (CP-868,596)
- Cohort C (Experimental): Adult patients with biopsy proven low grade glioma who have residual measurable disease. Patients are treated with Crenolanib (CP-868,596) continuously until they fulfill one of the criteria for study discontinuation.
  Interventions: Drug: Crenolanib (CP-868,596)

INTERVENTIONS:
Drug: Crenolanib (CP-868,596) — Highly potent inhibitor of both PDGFR receptors alpha and beta
  Other Names: Crenolanib Besylate

SUMMARY:
The purpose of this study is to evaluate the antitumor efficacy of crenolanib (CP-868,596) in patients with recurrent high grade glioma and in patients with low grade glioma.

DETAILED DESCRIPTION:
This Phase II study is designed to evaluate the antitumor efficacy of crenolanib (CP-868,596) in patients with recurrent high grade glioma and in patients with low grade glioma. Concurrently, the pharmacokinetics, tumor penetration and ability of crenolanib (CP-868,596) to inhibit PDGFR signaling will be evaluated when given as neo-adjuvant therapy to patients with radiographic evidence of malignant glioma prior to initial surgery.

The study will enroll 3 different cohorts of patients in parallel. Cohort A will enroll patients scheduled to undergo craniotomy and resection of newly diagnosed gliomas (both low and high grade). Patients in cohort A will be treated with crenolanib (CP-868,596) (300mg once daily, on an empty stomach) in the neo-adjuvant setting for a minimum of 3 days prior to surgical resection of their tumor mass. Twelve patients will be accrued on this neo-adjuvant cohort that will allow us to assess the ability of crenolanib (CP-868,596) to penetrate the tumor, not only in grade 3 and 4 gliomas (anaplastic astrocytomas and glioblastomas) that have a leaky BBB, but also in grade 2 gliomas (low grade gliomas) that tend to have a more intact blood-brain barrier (BBB).

Pharmacokinetic, pharmacodynamic and biological assessments will be conducted with tissue samples (plasma and brain tissue) obtained from these patients, when feasible.

Cohorts B and C will enroll patients with recurrent high grade gliomas or biopsy proven low grade glioma, respectively, who have residual measurable disease. Patients in cohorts B and C will be treated with crenolanib (CP-868,596) (300mg once daily on an empty stomach) continuously until they fulfill one of the criteria for study discontinuation. Magnetic resonance imaging (MRI) will be done to assess the tumor response as well as progression free survival (PFS). The primary endpoint for both cohorts B and C will be overall response rate according to the Response Evaluation Criteria In Solid Tumors (RECIST), as assessed by standard imaging modalities. In addition, 6-month Progression-free survival (cohort B) and 1-year PFS will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any racial or ethnic group
* Age 18 years or older
* Patient able and willing to provide informed consent
* Adequate kidney and liver function
* Karnofsky Performance Status ≥ 70%
* Negative serum pregnancy test or child bearing potential terminated by surgery, radiation, menopause or current use of two approved methods of birth control
* Imaging suggestive of malignant glioma (Cohort A)
* History of glioma with measurable disease by MRI (Cohorts B and C)
* Histologically confirmed GBM with radiographic progression (Cohort B). These patients are permitted to have had prior therapy including surgery, radiation, Temozolomide, irinotecan and bevacizumab.
* Histological confirmation of a low-grade glioma (Cohort C)

Exclusion Criteria:

* Patient unable to provide informed consent (comatose or markedly cognitively impaired)
* Female participants that are pregnant or breastfeeding
* Any other concurrent anticancer therapy
* Karnofsky Performance status < 70%
* Any other concurrent investigational agents within 4 weeks of start of study drug
* Patients with liver disease (known or active Hepatitis B or C; steatohepatitis; cirrhosis)
* Hepatic:

  * Bilirubin greater than 1x the upper limit of normal
  * Transaminases greater than 1x the upper limit of normal
* Abnormal renal function

  o Serum creatinine >1.7 ng/dl
* Patients on concomitant medications that induce or inhibit CYP450, such as enzyme inducing anti-epileptic drugs (EIAEDs) (Appendix III) and troglitazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary end-point is overall response rate | Tumor response will be assessed by MRI scans every 2 months until disease progression

SECONDARY OUTCOMES:
The secondary end-point for this study is PFS | 6-months and 12-months PFS will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Maher, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Harold Simmons Comprehensive Cancer Center, University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elizabeth A. Maher1, Clinton Stewart2, Kimmo Hatanpaa1, Jack Raisanen1, Tomoyuki Mashimo1, Xiao-Li Yang1, Chaitanya Muralidhara3, Christopher Madden1, Abhijit Ramachandran3, Bruce Mickey1, Robert Bachoo1, 1University of Texas Southwestern Medical Center, Dallas, TX, 2St. Jude's Children's Research Hospital, Memphis, TN, 3AROG Pharmaceuticals, LLC, Dallas, TX Neoadjuvant administration of the potent PDGFR inhibitor, crenolanib, to malignant gliomas at initial diagnosis: does it hit the target?
- See also: Harold C. Simmons Cancer Center at UT Southwestern is the only NCI-designated Cancer Center in North Texas — http://www.simmonscancercenter.org/index.html